CLINICAL TRIAL: NCT02761395
Title: Study of The Therapeutic Benefits of Al-hijamah in Children With Beta Thalassemia Major
Acronym: Al-hijamah
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2814/10/14
Record Dates: First submitted 2016-01-30; First posted 2016-05-04 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2016-04

CONDITIONS: AL-Hijama in Thalassmia Major
MeSH Terms: interventions — Deferasirox

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: ALhijama (Experimental): 20 patients under went Al-hijamah procedure for iron chelation
  Interventions: Procedure: Al-hijamah
- Group 2: AL-hijama with deferasirox (Experimental): 20 patients receive deferasirox and Al-hijamah.
  Interventions: Procedure: Al-hijamah; Drug: Deferasirox
- Group 3:deferasirox (Active Comparator): 20 patients already receiving deferasirox
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Procedure: Al-hijamah — * Strict sterilization of selected anatomical sites.
  * Suction using sterile plastic disposable sucking cups
  * Skin scarifications (shartat mihjam): through inducing superficial (0.1 mm in depth), small (2 mm in length), multiple and evenly distributed skin incisions.
  Arms: Group 1: ALhijama; Group 2: AL-hijama with deferasirox
Drug: Deferasirox — 20-40 mg/kg/day orally
  Arms: Group 2: AL-hijama with deferasirox; Group 3:deferasirox

SUMMARY:
1. Evaluate the therapeutic effects, health benefits, and immunological effect of Al-hijamah in children with beta thalassemia major.
2. Evaluate the extent of clinical improvement, reductions in serum iron and ferritin, antioxidant status, in those patients.

DETAILED DESCRIPTION:
The present study will be carried on 60 children patients with β- thalassemia major attending The Hematology Unit of Paediatric Departments at Tanta University Hospital. Participants will divide into 3 groups:

Group 1: 20 patients receive Al-hijamah.

Group 2: 20 patients receive Al-hijamah plus iron chelation therapy.

Group 3: 20 patients receive iron chelation therapy only

Participants undergo:

1. Laboratory investigations:

   * CBC (complete blood count) of peripheral venous blood before Al-hijamah and daily after it.
   * Differences between CBC from venous blood and cupped blood (bloody excretion collected inside suction cups). Cupped blood is collected in heparin coated with and added to suction cups put on the skin surface.

     • Serum iron and ferritin before Al-hijamah and after it.

     • Serum iron and ferritin in cupped blood vs venous blood.

     • Serum lipid profile and glycosylated hemoglobin before Al-hijamah and after it.
     * Total antioxidant capacity and some serum oxidants e.g. malondialdehyde before and after treatment
     * Flow cytometric analysis of number of Natural killer cells, CD4 T helper cells and CD4/CD8 cells (optional) (cluster of differentiation). They were reported to improve markedly after Al-hijamah.
     * Estimating serum LDH, pyruvate (antioxidant) and lactate (metabolite of pyruvate through LDH) in thalassemia patients before and after Al-hijamah
2. Assessment of heart function by Echocardiographic study (before and 3 month after Al-hijamah):

   * lines of therapy:

Technical steps of Al-hijamah (Necessary equipments are ready and can do it for all patients if possible):

Al-hijamah (Triple S technique under strict sterilization):

* Strict sterilization of selected anatomical sites.
* Suction using sterile plastic disposable sucking cups
* Skin scarifications (shartat mihjam): through inducing superficial (0.1 mm in depth), small (2 mm in length), multiple and evenly distributed skin incisions.
* Suction using sterile plastic disposable sucking cups
* Strict sterilization of selected anatomical sites.

Study endpoint:

This study will be terminated if safety of the patient were in dangers due to elements related to the new therapeutic agent or if the treatment not proven efficacious.

5. Risks to participants are reasonable in relation to anticipated benefits. Many human studies have proven safety of Al-hijamah.

6. Compensations of controls for transportation or work absence and of patients for any injury, and if so, description of the compensation should be mentioned.

No, compensations.

7. The proposal include a clear statement that an informed consent will be obtained from all participants in this research.

ELIGIBILITY:
Inclusion Criteria:

* Children suffering from beta thalassemia major, with age range from 4-18 years.

Exclusion Criteria:

* Children with Congenital heart disease
* Children with Rheumatic heart disease
* Presence of heart failure
* Children with Coronary arterial disease
* Children with Cardiomyopathy
* Children with hypotension
* Children with inflammatory skin diseases e.g. acute burns

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
CD(cluster of differentiation)4 and CD8 count | 3month
  count and percentage

SECONDARY OUTCOMES:
serum levels of cholesterol and triglyceride | 3month
  level of cholesterol and triglyceride (mg per dl)
alanine amino transferase , aspartate amino transferase | 3month
  measured as unit per litre
serum ferritin | 3 months
  measured as ng per dl
malodialdehyde ant total antioxidant capacity | 3 months
  measuedas mmol per litre

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed ELshanshory, prof, Study Director — ethical committee
Locations (1):
- Faculty of Medicine- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided